CLINICAL TRIAL: NCT05410769
Title: Compassionate Mind Training for Parkinson Patients and Caregivers
Brief Title: Compassion Program for Parkinson
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Nicola Modugno, Principal Investigator, Neuromed IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Compassion Focused Therapy
Record Dates: First submitted 2022-02-17; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD patients (Experimental): The intervention envisaged by the study takes place in the form of interviews, self-reports, and measurement of the heart rate variability.
  Interventions: Behavioral: Compassion Focused Therapy
- patient's caregivers (Experimental): The intervention envisaged by the study takes place in the form of interviews, self-reports, and measurement of the heart rate variability.
  Interventions: Behavioral: Compassion Focused Therapy

INTERVENTIONS:
Behavioral: Compassion Focused Therapy — This pilot study aims to propose for the first time a Compassion protocol (Compassion Program for Parkinson) to a group of patients with PD and a group of caregivers and to evaluate its feasibility and effectiveness. The investigators aim to assess whether the program is effective in improving the quality of life and psychiatric symptoms of the patients and caregivers. The Compassion program is a healthy form of self- acceptance, which involves being touched by one's own suffering, along with the desire to alleviate it and treat oneself with understanding and kindness. The duration of the protocol will be 6 weeks (1 meeting/ week of 2 hours). The investigators will recruit 40 patients and 20 caregivers who will be assessed pre and post intervention (Compassionate Mind Training) with interviews, self reports and measurement of the heart rate variability.

SUMMARY:
Parkinson's disease (PD) is a chronic and progressive neurodegenerative disease of the central nervous system. Second only to Alzheimer's in incidence on the population, Parkinson's disease has a negative impact on the quality of life of both patients and caregivers. Despite the prevailing attention to motor symptoms, such as bradykinesia, tremor and rigidity, the typical Parkinsonian symptom includes a wide range of non-motor symptoms that invalidate various aspects of the patient's autonomy, cognitive, behavior and mood that impact on patients' quality of life and that of caregivers.

DETAILED DESCRIPTION:
Non-motor symptoms in Parkinson's disease are classified in sensory, autonomic, behavioral, cognitive, sleep and psychic disorders. The most frequently presented neuropsychiatric symptoms are anxiety, depression, apathy, and impulsivity.

Although there are many false beliefs that patients often construct about their disease, PD patients still maintain a certain lucidity throughout the duration of the disease and its degeneration, improving the anxious-depressive symptoms. Psychic disorders can affect the patient's awareness of self-efficacy and self-regulation, as well as decision making capacity, mechanisms connected with dopaminergic circuits, the main target of PD neurodegeneration.

Parallel to the onset of symptoms in the patient, there is a great involvement of the caregivers who, aggravated by the emotional and welfare burden, develop over time stress, burden and burnout syndromes. The quality of life of caregivers undergo an objective impoverishment attributable to the inevitable alterations of free time and social relationships, in addition to a clinical psychophysical outcome.

Although there are numerous effective pharmaco-therapeutic approaches for motor symptoms, still little attention is paid to the prevention and treatment of neuropsychiatric symptoms.

Although there are still few studies, a new perspective of integrated care has gain attention due to the advantage of being able to be adapted to the needs and characteristics of the individual patient, enabling to choose the complementary / integrated therapy modality that best suits personal needs.

Within psychology, mindfulness practices such as MBSR Mindfulness protocols for stress have been successfully applied in different settings and on both patients and caregivers.

In the last twenty years, Compassion Focused Therapy practices increased within clinical practice, proving to be an adequate tool for improving psychophysical well-being. Compassion derives from the attachment behavioral system typical of mammals and allows the regulation of basic emotional systems. Compassion is divided into three streams: compassion towards oneself (Self-Compassion), compassion towards others and received from others. In particular, training one's Self Compassion through a Compassionate Mind Training can lead to proactive behaviors that improve the quality of one's life rather than enduring in a condition of passivity. Scientific research shows reliable data on the fact that awareness and compassion practices have physiological as well as psychological effects, acting on digestion, blood pressure, interbeat variability, but also on neuronal circuits. Recent studies correlate the levels of Compassion with a variation in HRV (heart rate variability) levels and has been suggested as a biomarker reliable in detecting the functions of the autonomic system. Variations in HRV values have been associated with autonomic dysfunctions, mood fluctuations and anxiety states in healthy subjects and subjects with generalized anxiety disorder.

Due to the persistent and still present pandemic emergency, the psychological symptoms are exacerbated by the general state of anxiety and uncertainty as well as by the inability to access public services. The conception of this "online study" is to allow a considerable possibility of interconnection and exchange, much easier in terms of technological means and timing.

This pilot study aims to propose for the first time an online Compassion (Compassion Program for Parkinson) protocol to a group of patients with PD and a group of caregivers and to evaluate its feasibility and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* PD diagnosis according to UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria (UKPDS)
* Ability to provide written informed consent
* Age between 18 and 80 years (inclusive)

Exclusion Criteria:

* cognitive impairment
* Inability to provide written informed consent
* any cardiological condition/drugs that alter the heartbeat
* Diagnosis of other concomitant neurodegenerative disease or psychiatric diaseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Compassion Mind Training online | 6 weeks
  Patients and Caregivers report on the Compassion Scale (Gilbert P. Compassion-focused therapy: Preface and introduction for special section. Br J Clin Psychol. 2014 Mar;53(1):1-5. doi: 10.1111/bjc.12045. PMID: 24588759.). CMT is a 6-session program, each lasting about 2 hours, which run on a weekly basis. The program is organized across 3 modules: 1) Our mind according to a compassion-based approach (to provide insight into the evolved and socially shaped mind and the affect regulation systems); 2) Compassionate mind training (understanding and cultivating the attributes and competencies of compassion in its three flows, and addressing its fears); and 3) final session (revising key information and practices and its application to the online routines).

SECONDARY OUTCOMES:
2. Beck Depression Inventory - II (BDI-II) | week 0, week 9, week 12
  Self-report questionnaire, depression symptom severity, scores can range from 0 to 63, with higher scores indicating more severe depression.
Change in quality of life | week 0, week 9, week 12
  Change from baseline in quality of life measured with the Parkinson Disease Questionnaire-39. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month covering 8 dimensions scored on a 5 point ordinal system (0=never, 4=always). Lower scores reflect better QoL.
Anxiety state | week 0, week 9, week 12
  The State-Trait Anxiety Inventory (STAI-Y) A which assessed the anxiety state (20 items; range, 20-80; < 35 = very low anxiety state, 36-45 = low anxiety state, 46-55 = medium anxiety state, 56-65 = high anxiety state, >65 = very high anxiety state).
Change from baseline in isolated heart rate variability at 12 weeks post CMT | week 0, week 9, week 12
  Pulse measurements at each online visit before and after the treatment period, At 3 time points during the online visit: 1-resting, 2-deep breathing, 3- post trigger interview.
  The incidence of clinically significant abonormal values will be summarized using descriptive statistics.

REFERENCES:
- [Background] Gilbert P. Compassion-focused therapy: Preface and introduction for special section. Br J Clin Psychol. 2014 Mar;53(1):1-5. doi: 10.1111/bjc.12045. No abstract available. PMID 24588759